CLINICAL TRIAL: NCT01494337
Title: Randomized Study Comparing Holmium Laser Enucleation of the Prostate (HOLEP) Versus Greenlight (XPS) Laser Photoselective Vapo-Enucleation of Prostate(PVEP) in the Management of Infravesical Obstruction Secondary to BPH
Brief Title: Holmium Laser Enucleation of Prostate(HOLEP) vs Greenlight(XPS) Laser Photoselective Vapo-Enucleation of Prostate(PVEP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royal Victoria Hospital, Canada (Other)
Collaborators: McGill University (Other)
Responsible Party: Principal Investigator, Mostafa Elhilali, clinical professor, Royal Victoria Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-171-SDR
Record Dates: First submitted 2011-12-05; First posted 2011-12-19 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Benign Prostate Hyperplasia
Keywords: LASER; BPH; Prostate surgery; HOLEP; Green light PVP
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HOLEP (Active Comparator): HOLEP In the first arm, holmium laser enucleation of the prostate will be done
  Interventions: Procedure: HOLEP
- PVEP/XPS (Active Comparator): PVEP/XPS green light photoselective Vapo-Enucleation of prostate using XPS 180W machine will be used in the second arm
  Interventions: Procedure: PVEP-XPS

INTERVENTIONS:
Procedure: HOLEP — USING HOLMIUM LASER, the prostate adenoma will be enucleated and removed into small pieces
  Other Names: Holmium Laser Enucleation of The Prostate
  Arms: HOLEP
Procedure: PVEP-XPS — Greenlight laser will be used with high power setting for selective vaporization of the prostate adenoma, using 180 watt XPS laser machine
  Other Names: Photoselective Vapo-Enucleation of prostate(PVEP)
  Arms: PVEP/XPS

SUMMARY:
The investigators are now proposing to compare two laser techniques for treating Benign prostate hyperplasia (BPH); Holmium Laser Enucleation of the Prostate (HOLEP) versus (greenlight) XPS which is a recently available technology in our center and is more efficient hence our choice to include patients with any size prostate. This will confirm whether the two techniques are equivalent in efficacy and safety independent of size as well as cost. The two techniques are available world wide as standard of care

DETAILED DESCRIPTION:
Patients with lower urinary tract symptoms (LUTS) secondary to bladder outlet obstruction from BPH seen through the outpatient clinic in the urology department will be assessed to see if the patient satisfies all inclusion and exclusion criteria. Patients who are meeting these criteria will be asked to participate in this randomized comparison study. If they agree they will be provided with an informed consent form which they can take home with them. The randomization process will be performed using computer-generated simple random tables in a 1:1 ratio. Study participants will be enrolled randomized, and the appropriate surgery scheduled. Procedures will be performed on an outpatient basis whenever possible.

All surgeries will be performed under a spinal or general anaesthesia. In case of coexisting vesical stone, Holmium laser cystolithotripsy will be done first regardless the type of next procedure for the prostate. Both HOLEP and greenLight (XPS) laser vaporization of the prostate begins with the insertion of a resectoscope transurethrally. Examination of the lower urinary tract is performed and holmium laser fiber is used to enucleate (HOLEP) or to vaporize [greenLight (XPS)] the obstructing prostatic tissue using the Moxy fibre until the surgical capsule is reached. After treatment, the prostatic fossa will be examined for hemostasis and if adequate, a 22 french Foley catheter will be inserted. Patients will then be sent to the post-anaesthetic recovery room.

Once awake, the patient could have the catheter removed with a voiding trial if the urine is judged to be sufficiently clear and the surgeon is comfortable about early catheter removal. Those patients able to void will be sent home without catheter. Those patients unable to void or the surgeon decides to keep the catheter for 24 hours will be either sent home with a catheter to be removed the next day or hospitalized overnight.

Finally, those patients with multiple medical problems or with postoperative bleeding requiring bladder irrigation will be kept overnight with a trial of voiding attempted the next morning if the urine is clear.

Intraoperative and early postoperative parameters of interest will be recorded and compared between groups. These parameters include the total procedure time, total laser energy used, cost of disposables including the number of laser fibers per case, number of bags of irrigant per case, urethral catheterization time, length of hospital stay, subjective assessment of hemostasis during each laser procedure, objective assessment of changes in serum electrolytes and hematocrit and thorough recording of all complications.

Patients will be seen in follow-up at 2 weeks, 1, 3, 6, and 12 months. The parameters to be assessed at each time point are listed below. As can be seen from the table, the most important parameters will be changes in voiding symptoms and uroflowmetry over time. Some validated questionnaires will be utilized to assess the patients' sexual function both at base line and at different follow-up visits. Different aspects of the sexual function will be analysed, partner's feedback will be addressed by a special questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent.
2. Lower urinary symptoms (LUTS) secondary to bladder outlet obstruction from BPH.
3. Failed medical treatment of BPH.
4. International prostate symptom scores (IPSS) > 15.
5. Peak urinary flow rate (Qmax) < 15 ml/sec.
6. Preoperative TRUS (transrectal ultrasound) size of the gland (from 40 to 150 cc).
7. Patients in retention secondary to BPH (with cystometrogram (CMG) confirming adequate detrusor pressure if the bladder capacity at time of catheterization is in excess of 1000 ml).

Exclusion Criteria:

1. Inability to give informed consent.
2. Patient who have a neurological disorder which might affect bladder function as cerebrovascular stroke, Parkinson disease.
3. Active urinary tract infection.
4. Presence of active bladder cancer (within the last 2 years).
5. Known cancer prostate patients will be excluded preoperatively on the basis of digital rectal examination, prostate specific antigen level, and TRUS imaging followed by prostate biopsies if necessary.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
change in urine flow parameters | one, 4 and 12 months postoperative
  change in urine flow parameters; IPSS= international prostate symptom score QOL= quality of life score PVR= post voiding residual urine Q-MAX= maximal flow rate

SECONDARY OUTCOMES:
TIME TO CATHETER REMOVAL, HOSPITAL STAY | 1 day post operative
  At first postoperative day; the catheter will be removed for trial voiding Patient will be discharged from the hospital as soon as possible (same day or once urine color is normalized)
the need for redo surgery | 1 year
  The need for re-operation in the fist year will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa M Elhilali, Professor, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Royal victoria hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Elshal AM, Elkoushy MA, El-Nahas AR, Shoma AM, Nabeeh A, Carrier S, Elhilali MM. GreenLight laser (XPS) photoselective vapo-enucleation versus holmium laser enucleation of the prostate for the treatment of symptomatic benign prostatic hyperplasia: a randomized controlled study. J Urol. 2015 Mar;193(3):927-34. doi: 10.1016/j.juro.2014.09.097. Epub 2014 Sep 28. PMID 25261801